CLINICAL TRIAL: NCT04756375
Title: Evaluation of Virtual Reality to Save Morphinic in the Treatment of Vaso-occlusive Seizures of Sickle Cell Patients Consulting in the Emergency Room
Acronym: ReVCVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP190729; IDRCB2020-A00599-30 (Other: ANSM)
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Vaso-occlusive Crisis; Sickle Cell Disease
Keywords: Virtual reality; Vaso occlusive seizure; Sickle Cell Disease; Emergency Room; Pain
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell; Emergencies; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): Use of virtual reality in the management of sickle cell patients with VOS
  Interventions: Device: Virtual Reality
- NO INTERVENTION (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Virtual Reality — Use of virtual reality in the management of sickle cell patients with VOS
  Arms: INTERVENTION
Other: Usual Care — Usual management of sickle cell patients with VOS
  Arms: NO INTERVENTION

SUMMARY:
The management of pain in the emergency department is a major issue, especially for sickle cell patients who regularly consult for vaso-occlusive seizure (VOS). The place of virtual reality remains to be defined in a busy environment, in which the permanence of care generates a significant turn over of medical and paramedical personnel.

With Its immersive nature, allowing the patient to detach from his immediate environment, wich is often stressful for patients, we can hope that in multimodal management, Virtual Reality (VR) can contribute to a faster reduction in pain with lower doses of morphine, but so far we have no data.

Our pilot study aims to assess the effectiveness, feasibility and tolerance of adding virtual reality to the management of VOS in sickle cell patients in the ER.

DETAILED DESCRIPTION:
It will be a Before-after study: this study will be conducted in 2 phases in the emergency department

* a period of usual management of sickle cell patients with VOS
* then a phase during which the device will be used. Each phase will last 3 months; the duration of the periods may be shorter if recruitment targets are met. Patients will be included consecutively.

The main objective of the study is to measure the impact of virtual reality on the total dose of morphine administered to the emergency room in the treatment of vaso-occlusive seizures after initial morphine titration.

The primary endpoint is the total dose of morphine (in milligrams), used in the emergency room after initial titration, meaning the dose administered by PCA (patient-controlled analgesia) and secondary titrations in the event of a recurrence of painful spikes with analog verbal scale (AVS) >7.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* sickle cell patient consulting in the emergency room for VOS
* Signature free and informed consent

Exclusion Criteria:

* Consultation in the ER for the same reason in the 14 days prior to inclusion (same episode)
* Emergency room consultation more than 12 times in the previous year
* Nausea and vomiting at the time of inclusion
* History of epilepsy
* A visually impaired or hard of hearing patient
* Pregnant patient
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine | up to 48 hours
  Total dose of morphine (in milligrams), used in the emergency room after initial titration, meaning the dose administered by PCA and secondary titrations in case of recurrence of painful peak with AVS>7

SECONDARY OUTCOMES:
Feasibility of implementing the scheme | up to 48 hours
  Number of patents included in the protocol vs. number of potentially eligible patients For patients included during the VR period: the number of VR sessions performed, and the duration of these sessions.
Tolerance | up to 48 hours
  Side effects such as headache, nausea, eye pain or dizziness
Acceptability | up to 48 hours
  Patient's willingness to use VR again at future VOS Evaluation of patient satisfaction
Pain Efficiency | up to 48 hours
  Evaluation of AVS before and after the virtual reality session Numbers of painful areas before and after virtual reality

CONTACTS AND LOCATIONS:
Overall Officials: Hélène GOULET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOPITAL TENON Service des urgences, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided